CLINICAL TRIAL: NCT02454101
Title: Milking Versus Delayed Cord Clamping in Full Term Neonates Delivered by Elective Cesarean Section A Randomized Controlled Trial
Brief Title: Milking Versus Delayed Cord Clamping in Full Term Neonates
Acronym: MDCCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Mohamed El Kotb Abdel Fattah (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: delayed cord clamping in term
Record Dates: First submitted 2015-05-17; First posted 2015-05-27 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-04

CONDITIONS: Neonatal Anemia
MeSH Terms: conditions — Anemia, Neonatal | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cord milking (Other): milking of the umbilical cord 5 times toward the neonate
  Interventions: Procedure: delayed cord clamping
- delayed cord clamping (Other): delayed cord clamping for 120 seconds
  Interventions: Procedure: cord milking

INTERVENTIONS:
Procedure: cord milking — milking of the cord 5 times toward the neonate
  Other Names: milking of the cord
  Arms: delayed cord clamping
Procedure: delayed cord clamping — delay clamping of the cord for 120 seconds
  Arms: cord milking

SUMMARY:
To compare the short term risks and benefits of cord milking 5 times toward the neonate with delayed cord clamping for 120 seconds in the full term neonate delivered by cesarean section.

DETAILED DESCRIPTION:
Abstract Context: milking of the umbilical cord toward the neonate 5 times and delayed cord clamping both are good procedures to prevent anemia in neonates .

Objective: To investigate the effects of delayed umbilical cord clamping for 120 seconds, compared with milking of the cord 5 times toward the neonate on hemoglobin level after 6 weeks, Intubation,Respiratory distress,Clinical jaundice,Neonatal Intensive Care unit (NICU) admission,Apgar score (after 5 minutes of delivery).

-Maternal,Need for blood transfusion,Additional need for therapeutic uterotonics,Post postpartum hemorrhage (blood loss > 500cc),Intensive Care unit admission.

Design: Randomized controlled trial. Setting: Ain Shams university maternity hospital. Participants:300 full term infants born after a low risk pregnancy by cesarean section delivery.

Intervention: Infants were randomized to delayed umbilical cord clamping (≥120 seconds after delivery) or cord milking (5 times to ward the neonate).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females going for cesarean section that completed 37 weeks of gestation
* Medically free

Exclusion Criteria:

* Known congenital anomalies of fetus.
* Rhesus sensitization.
* Fetal hydrops.
* Medical disorder (preeclampsia - diabetes mellitus - hypertension - SLE).
* Need for urgent resuscitation.
* Multiple pregnancies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hazem F El Shahawy, PHD, Principal Investigator — clinical professor
Locations (1):
- Ain Chams University Maternity Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
lecture and seminar

REFERENCES:
- [Background] Carlson ES, Tkac I, Magid R, O'Connor MB, Andrews NC, Schallert T, Gunshin H, Georgieff MK, Petryk A. Iron is essential for neuron development and memory function in mouse hippocampus. J Nutr. 2009 Apr;139(4):672-9. doi: 10.3945/jn.108.096354. Epub 2009 Feb 11. PMID 19211831
- [Background] Chaparro CM, Neufeld LM, Tena Alavez G, Eguia-Liz Cedillo R, Dewey KG. Effect of timing of umbilical cord clamping on iron status in Mexican infants: a randomised controlled trial. Lancet. 2006 Jun 17;367(9527):1997-2004. doi: 10.1016/S0140-6736(06)68889-2. PMID 16782490
- [Background] Eichenbaum-Pikser G, Zasloff JS. Delayed clamping of the umbilical cord: a review with implications for practice. J Midwifery Womens Health. 2009 Jul-Aug;54(4):321-6. doi: 10.1016/j.jmwh.2008.12.012. No abstract available. PMID 19555916
- [Background] Emhamed MO, van Rheenen P, Brabin BJ. The early effects of delayed cord clamping in term infants born to Libyan mothers. Trop Doct. 2004 Oct;34(4):218-22. doi: 10.1177/004947550403400410. PMID 15510946
- [Background] Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. doi: 10.1001/jama.297.11.1241. PMID 17374818
- [Background] Inch S. Management of the third stage of labour: another cascade of intervention?. Midwifery 1985;1:114-22.
- [Background] Ladipo OA. Management of third stage of labour, with particular reference to reduction of feto-maternal transfusion. Br Med J. 1972 Mar 18;1(5802):721-3. doi: 10.1136/bmj.1.5802.721. PMID 5015327
- [Background] McCann JC, Ames BN. An overview of evidence for a causal relation between iron deficiency during development and deficits in cognitive or behavioral function. Am J Clin Nutr. 2007 Apr;85(4):931-45. doi: 10.1093/ajcn/85.4.931. PMID 17413089
- [Background] .McDonald S. Physiology and management of the third stage of labour. In: Fraser D, Cooper M editor(s). Myles textbook for mid- wives. 14th Edition. Edinburgh: Churchill Livingstone, 2003.
- [Background] Mercer JS. Current best evidence: a review of the literature on umbilical cord clamping. J Midwifery Womens Health. 2001 Nov-Dec;46(6):402-14. doi: 10.1016/s1526-9523(01)00196-9. PMID 11783688
- [Background] .Prendiville W, Elbourne D. Care during the third stage of labour. In: Chalmers I, Enkin M, Keirse MJNC editor(s). Effective care in pregnancy and childbirth. Oxford: Oxford University Press, 1989: 1145-69.
- [Background] Rabe H, Reynolds G, Diaz-Rossello J. Early versus delayed umbilical cord clamping in preterm infants. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003248. doi: 10.1002/14651858.CD003248.pub2. PMID 15495045
- [Background] Rabe H, Reynolds G, Diaz-Rossello J. A systematic review and meta-analysis of a brief delay in clamping the umbilical cord of preterm infants. Neonatology. 2008;93(2):138-44. doi: 10.1159/000108764. Epub 2007 Sep 21. PMID 17890882
- [Background] .Smith J, Brennan BG. Management of the third stage of labor. EMedicine from WebMD (last updated 27 June 2006) (accessed 28 January 2007).
- [Background] Szajewska H, Ruszczynski M, Chmielewska A. Effects of iron supplementation in nonanemic pregnant women, infants, and young children on the mental performance and psychomotor development of children: a systematic review of randomized controlled trials. Am J Clin Nutr. 2010 Jun;91(6):1684-90. doi: 10.3945/ajcn.2010.29191. Epub 2010 Apr 21. PMID 20410098
- [Background] Thane CW, Walmsley CM, Bates CJ, Prentice A, Cole TJ. Risk factors for poor iron status in British toddlers: further analysis of data from the National Diet and Nutrition Survey of children aged 1.5-4.5 years. Public Health Nutr. 2000 Dec;3(4):433-40. doi: 10.1017/s1368980000000501. PMID 11135798
- [Background] Thomas DG, Grant SL, Aubuchon-Endsley NL. The role of iron in neurocognitive development. Dev Neuropsychol. 2009;34(2):196-222. doi: 10.1080/87565640802646767. PMID 19267295
- [Background] van Rheenen PF, Brabin BJ. A practical approach to timing cord clamping in resource poor settings. BMJ. 2006 Nov 4;333(7575):954-8. doi: 10.1136/bmj.39002.389236.BE. No abstract available. PMID 17082547
- [Background] Yao AC, Lind J. Placental transfusion. Am J Dis Child. 1974 Jan;127(1):128-41. doi: 10.1001/archpedi.1974.02110200130021. No abstract available. PMID 4588934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The current RCT was conducted at Ain Shams University Maternity Hospital during the period between August 2015 to February 2016
Pre-assignment Details: No significant events following participants recruitment
Period: Overall Study
Arm/Group | Cord Milking | Delayed Cord Clamping
Started | 150 | 150
Completed | 145 | 143
Not Completed | 5 | 7
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cord Milking | Delayed Cord Clamping | Total
Number analyzed (Participants) | 145 | 143 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.42 (1.67) | 22.4 (1.78) | 22.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 143 | 288
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 145 | 143 | 288

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Hemoglobin Level
Description: neonatal 6 weeks hemoglobin measured in gram %
Time Frame: 6 weeks after labor
Population: Number of Infants Analyzed
Measure: Mean (Standard Deviation); unit: gram%
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
gram% | 11.86 (0.71) | 11.95 (0.88)

2. Secondary Outcome: Jundice Requring Phtotherapy
Description: number of infants requiring phtotherapy for jundice in the first 2 weeks
Time Frame: two weks
Population: Number of Infants Analyzed
Measure: Number; unit: participants
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
participants | 16 | 12

3. Secondary Outcome: Severe Postpartum Haemorrage
Description: (measured blood loss 1000 mL or more
Time Frame: 24 hours after labor
Measure: Number; unit: participants
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
participants | 4 | 2

4. Secondary Outcome: Neonatal Intubation
Description: number of newborns requirng intubation in the first 2 hours after delivery
Time Frame: 1st 2 hours after delivery
Population: Number of Infants Analyzed
Measure: Number; unit: participants
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
participants | 0 | 0

5. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission
Description: number of Neonatal Intensive Care unit (NICU) admission in the 1st 24 hours after delivery
Time Frame: 1st 24 hours after delivery
Population: Number of Infants Analyzed
Measure: Number; unit: participants
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
participants | 17 | 15

6. Secondary Outcome: Neonatal Apgar Score (After 5 Minutes of Delivery).
Description: * The Apgar test is done by a doctor, midwife, or nurse. The health care provider examines the baby's:
    1. Breathing effort
    2. Heart rate
    3. Muscle tone
    4. Reflexes
    5. Skin color
  * Each category is scored with 0, 1, or 2, depending on the observed condition.
  * The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth.
  * A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health. A score of 10 is very unusual, since almost all newborns lose 1 point for blue hands and feet, which is normal for after birth.
  * Any score lower than 7 is a sign that the baby needs medical attention. The lower the score, the more help the baby needs
Time Frame: 5 minutes of delivery
Population: Number of Infants Analyzed
Measure: Mean (Standard Deviation); unit: Scores on a Scale from 1 to 10
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
Scores on a Scale from 1 to 10 | 8.73 (0.58) | 8.26 (0.66)

7. Secondary Outcome: Maternal Need for Blood Transfusion.
Description: number of mothers with hemoglobin level < 7mg/dl and need for blood transfusion
Time Frame: 1st 24 hours after delivery
Measure: Number; unit: participants
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
participants | 1 | 2

8. Secondary Outcome: Maternal Additional Need for Therapeutic Uterotonics
Description: number of mothers need for > 20 units of Oxycontin in the 1st 24 hours of delivery
Time Frame: 1st 24 hours of delivery
Measure: Number; unit: participants
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
participants | 8 | 10

9. Secondary Outcome: Duration of Third Stage of Labor
Description: number of minutes from delivery of the baby till delivery of the placenta
Time Frame: immediatly after delivery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cord Milking | Delayed Cord Clamping
Number analyzed (Participants) | 145 | 143
minutes | 5.45 (2.56) | 8.56 (3.15)

ADVERSE EVENTS:
Time Frame: 6 MONTHS
Description: Postpartum haemorrage defined as loss of more than 1000 ml blood during the first 24 hours after delivery
Arm/Group | Cord Milking | Delayed Cord Clamping
Serious Adverse Events (participants affected / at risk) | 4/145 | 2/143
Other Adverse Events (participants affected / at risk) | 12/145 | 14/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cord Milking (N=145) | Delayed Cord Clamping (N=143)
post partum haemorrage (Blood and lymphatic system disorders) | 4 (4) | 2 (2) — loss of more than 1000 ml of blood after delivery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cord Milking (N=145) | Delayed Cord Clamping (N=143)
need for blood trasnfusion (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Need for manual Removal of the placenta (Surgical and medical procedures) | 3 (3) | 2 (2)
Need for Therapeutic Uterotonics (Surgical and medical procedures) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No